CLINICAL TRIAL: NCT07144540
Title: The Effectiveness of NeuroBot in Alleviating Anxiety of Patients Undergoing Neurovascular Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other); Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, HO Chung Man, Doctor of Nursing Student, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NeuroBot202527
Record Dates: First submitted 2025-08-15; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Patient Compliance; Knowledge
Keywords: Chatbot; NeuroBot; Perioperative education; Neurovascular surgery
MeSH Terms: conditions — Anxiety Disorders; Patient Compliance | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The control arm will receive standard preoperative education in the preoperative nurse clinic, apart from face-to-face consultation, leaflet will be provided for illustrating the surgical procedure and the disease. For the intervention arm, on top of the standard care as above, they will be additionally provided an artificial intelligence chatbot "NeuroBot" for perioperative support.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care arm (Active Comparator): The participants will receive standard perioperative care as usual care
  Interventions: Other: Standard Care (in control arm)
- NeuroBot arm (Experimental): Patients will receive additional support from NeuroBot during perioperative period
  Interventions: Other: NeuroBot; Other: Standard Care (in control arm)

INTERVENTIONS:
Other: NeuroBot — NeuroBot is an artificial intelligence online accessible chatbot that used machine learning and generative pretrained transformer model for supporting patients undergoing neurovascular surgery during perioperative period
  Arms: NeuroBot arm
Other: Standard Care (in control arm) — Standard care include face-to-face consultation in preoperative nurse clinic and provision of leaflet

SUMMARY:
The goal of this randomized controlled trial is to investigate the effectiveness of NeuroBot in alleviating anxiety of patients undergoing neurovascular procedures. The main questions it aims to answer are:

Is NeuroBot effective in alleviating anxiety? Is NeuroBot effective in enhancing patients' procedure and disease-related knowledge? Is NeuroBot effective in enhancing patients' compliance to treatment? If there is a comparison group: Researchers will compare with standard perioperative education (control group) to see if there is any difference in results.

Participants will be invited to chat with the artificial intelligence based chatbot "NeuroBot" for 6 weeks, from the date of preoperative clinic visit till 4 weeks after the surgery. The participants are allowed to access the NeuroBot at anytime anywhere, to ask surgery- related questions at their discretion.

DETAILED DESCRIPTION:
The NeuroBot is co-developed by the neurosurgeons, nuerosurgical specialty nurses in Queen Elisabeth Hospital and AI experts from the Hong Kong Polytechnic University and the Chinese University of Hong Kong. The NeuroBot is developed based on the large language model that used machine learning algorithm and generative pretrained transformer model. Vast dataset of neurovascular surgery related information from validated sources, including DynaMed, UpToDate and textbooks were included and used for training of NeuroBot. The precision of the responses generated by NeuroBot was verified by a group of neurosurgical domain experts (neurosurgeons and experienced neurosurgical nurses).

ELIGIBILITY:
Inclusion Criteria:

1. aged above 18 years;
2. scheduled for elective neuroendovascular surgery;
3. able to understand Chinese and read Chinese;
4. mobile device with internet capability.

Exclusion Criteria:

1. identified cognitive impairment or have difficulty in understanding study procedures, following instructions, or providing informed consent;
2. prior exposure to health chatbot to acquire health-related information in previous 3 months;
3. have neurovascular surgeries before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From preoperative (at nurse clinic) to postoperative from 1 week to 4 weeks after surgery
  Level of preoperative and postoperative anxiety, measured using State Trait Anxiety Inventory - State scale (6-item Chinese version). There are total of 6-item in the questionnaire, each item uses a 1 to 4 point rating scale. 1: not at all; 2: somewhat; 3: moderate; 4: very much so. The higher the score indicates the greater levels of anxiety

SECONDARY OUTCOMES:
Knowledge | From preoperative nurse clinic visit to 1 week postoperative
  The level of procedure and disease related knowledge. A 10-item multiple choice questionnaire was developed and validated by neurosurgical experts. It will be used to assess participants' level of knowledge. Each participant will score 1 mark if they correctly answer each question. The higher the score, the higher the level of knowledge.
Compliance | 4 weeks after surgery
  Compliance to prescribed treatment including follow-up visit, arranged investigation. The incidence of non-compliance will be traced through reviewing medical records. Each missed follow-up visit and investigation within 1 month after surgery will be counted. Each incidence of missed follow-up visits and investigations will be descriptively reported in both groups
Readmission | 4 weeks after surgery
  Readmission related to the surgery. The incidence of readmission related to the postoperative complications will be traced in medical record. Number of Participants with readmission will be descriptively reported.
Postoperative complications | 4 weeks after surgery
  surgery-related postoperative complications. The incidence of surgery-related postoperative complications will be traced in medical record. Number of Participants with surgery-related postoperative complications will be descriptively reported in both groups

OTHER OUTCOMES:
Perception on the usability of NeuroBot | 4 weeks after surgery
  Conduct qualitative interview for a group of participants in the intervention group to evaluate the usefulness of and satisfaction to the NeuroBot

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No